CLINICAL TRIAL: NCT06702332
Title: A Randomized, Double-blind, Placebo-controlled, Sequential, Adaptive Single Ascending Dose Study to Evaluate the Safety and Tolerability, Pharmacokinetics and Pharmacodynamic Profile of Orally Administered MSD-001 in Healthy Participants.
Brief Title: Single Ascending Dose Study of MSD-001 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mindstate Design Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSD001-NL-001; 2024-512939-67-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-11; First posted 2024-11-22 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-01

CONDITIONS: Mental Health Disorders

STUDY DESIGN:
Intervention Model Description: In Part 1, Participants (n=8) will be randomized to receive either MSD-001 or placebo (6 active: 2 placebo) in each of 5 ascending dose levels (cohorts).
  In Part 2, Participants (n=4) with a CYP2D6 poor metabolizing phenotype will all receive MSD-001 (4 active: 0 placebo) in each of 3 ascending dose levels (cohorts).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Treatment: MSD-001 (Active Comparator): Planned doses of MSD-001; N = 42
  Interventions: Drug: MSD-001
- Placebo Comparator (Placebo Comparator): Non-active study drug N = 10
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: MSD-001 — MSD-001 is being developed as part of future two-agent combination treatment approaches for the management of mental health indications
  Arms: Active Treatment: MSD-001
Drug: Placebo Comparator — Matching Placebo
  Arms: Placebo Comparator

SUMMARY:
The purpose of this Phase 1 single ascending dose (SAD) study is to evaluate the safety and tolerability, pharmacokinetics, and pharmacodynamic profile of MSD-001 when administered orally to healthy adult participants.

DETAILED DESCRIPTION:
This is a first in human, prospective, single center, double blind, placebo-controlled, single ascending dose study to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of MSD-001. The study will include two parallel parts, Part 1 and Part 2, stratified by CYP2D6 phenotype.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female healthy consented participants 18 to 55 years of age
* CYP2D6 phenotype established based on pharmacogenetic testing.
* Free from psychoactive drug use from 4 weeks before dosing and until the last follow up visit.

Key Exclusion Criteria:

* Any current clinically relevant, or history of, acute or chronic diseases inclusive of psychiatric disorders and relevant family history, which could interfere with the participant's safety during the trial, or expose them to undue risk, or which could interfere with the study objectives.
* Moderate to severe congestive heart failure, history of heart surgery, pulmonary hypertension, systemic hypertension (i.e., systolic BP >139 mm hg, diastolic blood pressure > 89 mm hg), pulse rate > 90 bpm, clinically significant ECG abnormality, QTc > 450 msec, myocardial infarction in the past year, or any other active or severe cardiovascular condition.
* Clinically significant personal or familial history of epilepsy, seizures, convulsions, or other seizure disorder (excluding febrile seizures as a child), previous head trauma or other risk factor for seizure.
* Use of any psychedelic drug in the three months prior to planned dosing or the occurrence of persistent psychological effects following the previous use of psychedelic drugs.
* Subject experiences severe anticipatory anxiety or is otherwise considered unfit for study.
* History of moderate or severe illicit substance abuse or dependence, or a positive test result(s) for alcohol and/or drugs of abuse at screening or admission to the clinical unit.
* Subject has received a prior investigational intervention, has had a history of relevant hypersensitivity or allergic reactions, and has donated and/or received any blood or blood products or experienced blood loss, that may interfere with the objectives of the study.
* Subject has a significant negative life event (e.g. loss of a loved one) in the past 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of MSD-001 in healthy adult participants by assessing the number, duration, severity, drug relatedness and type of adverse events | up to 30 days
  Treatment emergent adverse events/ treatment emergent serious adverse events - their frequency, duration and severity, clinically significant changes in lab parameters, ECG, and vital signs

SECONDARY OUTCOMES:
Plasma Pharmacokinetics (PK) of a single dose of MSD-001: Maximum Plasma Concentration (Cmax) | Pre-dose and up to 24 hours post dose
  Following completion of each cohort, bioanalytical analysis for MSD-001 serial PK timepoints will be performed and plasma PK parameters for Cmax analyzed
Plasma Pharmacokinetics (PK) of a single dose of MSD-001: time to attain Cmax (Tmax) | Pre-dose and up to 24 hours post dose
  Following completion of each cohort, bioanalytical analysis for MSD-001 serial PK will be performed and plasma PK parameters for Tmax analyzed
Plasma Pharmacokinetics (PK) of a single dose of MSD-001: Area under plasma Concentration (AUC) | Pre-dose and up to 24 hours post dose
  Following completion of each cohort, bioanalytical analysis for MSD-001 serial PK timepoints will be performed and plasma PK parameters for AUC analyzed
Plasma Pharmacokinetics (PK) of a single dose of MSD-001: terminal elimination half-life (T1/2) | Pre-dose and up to 24 hours post dose
  Following completion of each cohort, bioanalytical analysis for MSD-001 serial PK will be performed and plasma PK parameters for T1/2 analyzed
5D-ASC (5 dimensional altered states of consciousness) rating scale (a 94-item VAS questionnaire) | Pre-dose and 24 hours post dose
  Participants will be asked to reflect on the previous days' subjective experience using 5D-ASC rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Jacobs, MD, PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, South Holland, Netherlands